CLINICAL TRIAL: NCT00265772
Title: Phase IV Study Comparing a Nutritional Anti-Inflammatory Treatment to Steroids for Pediatric Crohn's Disease - the Molecular Basis
Brief Title: Comparison of a Nutritional Anti-Inflammatory Treatment to Steroids for Pediatric Crohn's Disease - the Molecular Basis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Société des Produits Nestlé (SPN) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCNF0105
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-11

CONDITIONS: Crohn's Disease; Pediatric
Keywords: enteral nutrition; steroids; mucosal healing
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Drug: MODULEN IBD (R) (specific Enteral Nutrition)
Drug: prednisolon

SUMMARY:
The primary purpose of this study is to compare the efficacy of enteral nutrition compared to steroids in inducing remission of active pediatric Crohn's disease. The main hypothesis of this study is that the use of enteral nutrition induces mucosal healing, whereas steroids do not. This effect may be related to a change of the commensal flora during enteral nutrition.

DETAILED DESCRIPTION:
The precise and exact cause of Crohn's disease (CD) remains still unknown. However, recent data point out to an inappropriate and exaggerated inflammatory response of the intestinal mucosal immune system toward intestinal commensal flora as initial trigger. Several strategies were developed in the treatment of active CD. Anti-inflammatory drugs such as steroids proved to be very helpful in the induction of a primary remission as is the use of exclusive enteral nutrition. Besides a long standing experience with EN in the management of CD in several centres, the mode of action and the molecular mechanisms of a specific EN, such as Modulen IBD ® remain still unknown. The ultimate aim of this study is to compare the efficacy of Modulen IBD ® in inducing remission compared to steroids with a detailed analysis of the mucosal repair and anti-bacterial defence mechanisms within the inflamed intestinal mucosa and the composition of the commensal flora before and during therapy. This approach may help to elucidate the interaction between the intestinal mucosa and the commensal flora during the onset of CD and induction of remission.

ELIGIBILITY:
Inclusion Criteria:

Crohn's disease active disease small bowel involvement

Exclusion Criteria:

antibiotic therapy within 4 weeks prior to inclusion immunosuppressive therapy within 4 weeks prior to inclusion not willing to collaborate isolated oral or perianal involvement

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24
Dates: Start 2005-11; Study Completion 2008-04

PRIMARY OUTCOMES:
Mucosal Healing (decrease >70% of the Crohn's disease endoscopic index score after 8 weeks of treatment)

SECONDARY OUTCOMES:
clinical remission (Harvey Bradshaw Index <5)
biological remission (decrease of systemic and mucosal inflammatory markers)
improvement of the anti-bacterial defense

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Ruemmele, MD PhD, Principal Investigator — Hôpital Necker Enfants Malades, Assistance Publique-Hôpitaux de Paris, Service de Gastroenterologie pédiatrique, INSERM EMI0212, Paris, France
Locations (1):
- Hôpital Necker Enfants Malades, Faculté de Médecine Necker, INSERM EMI0212, Paris, France

REFERENCES:
- [Background] Bannerjee K, Camacho-Hubner C, Babinska K, Dryhurst KM, Edwards R, Savage MO, Sanderson IR, Croft NM. Anti-inflammatory and growth-stimulating effects precede nutritional restitution during enteral feeding in Crohn disease. J Pediatr Gastroenterol Nutr. 2004 Mar;38(3):270-5. doi: 10.1097/00005176-200403000-00007. PMID 15076624
- [Background] Heuschkel RB, Menache CC, Megerian JT, Baird AE. Enteral nutrition and corticosteroids in the treatment of acute Crohn's disease in children. J Pediatr Gastroenterol Nutr. 2000 Jul;31(1):8-15. doi: 10.1097/00005176-200007000-00005. PMID 10896064
- [Background] Heuschkel RB, MacDonald TT, Monteleone G, Bajaj-Elliott M, Smith JA, Pender SL. Imbalance of stromelysin-1 and TIMP-1 in the mucosal lesions of children with inflammatory bowel disease. Gut. 2000 Jul;47(1):57-62. doi: 10.1136/gut.47.1.57. PMID 10861265
- [Background] Belli DC, Seidman E, Bouthillier L, Weber AM, Roy CC, Pletincx M, Beaulieu M, Morin CL. Chronic intermittent elemental diet improves growth failure in children with Crohn's disease. Gastroenterology. 1988 Mar;94(3):603-10. doi: 10.1016/0016-5085(88)90230-2. PMID 3123302
- [Background] Ruemmele FM, Roy CC, Levy E, Seidman EG. Nutrition as primary therapy in pediatric Crohn's disease: fact or fantasy? J Pediatr. 2000 Mar;136(3):285-91. doi: 10.1067/mpd.2000.104537. No abstract available. PMID 10700682
- [Background] Gailhoustet L, Goulet O, Cachin N, Schmitz J. [Study of psychological repercussions of 2 modes of treatment of adolescents with Crohn's disease]. Arch Pediatr. 2002 Feb;9(2):110-6. doi: 10.1016/s0929-693x(01)00717-5. French. PMID 11915490